CLINICAL TRIAL: NCT05106426
Title: Healthy Caregivers-Healthy Children Phase 3: Children With Special Needs
Brief Title: Healthy Caregivers-Healthy Children
Acronym: HC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ruby Natale, Associate Professor of Clinical Pediatrics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20210902
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Obesity; Child, Only
Keywords: obesity prevention; childhood; special needs
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HC2 intervention Group (Experimental): Participants in this group will receive the Healthy Caregivers-Healthy Children (HC2) intervention for 24 months
  Interventions: Behavioral: Healthy Caregivers- Healthy children
- Jump Start Control Group (Active Comparator): Participants in this group will receive the Jump Start intervention for 24 months
  Interventions: Behavioral: Jump Start
- Parents/Caregivers of Participants receiving HC2 intervention (No Intervention): Parents/caregivers of participants receiving the HC2 program will not be receiving any intervention.
- No Intervention: Parents/Caregivers of participants receiving Jump Start Intervention (No Intervention): Parents/caregivers of participants receiving the Jump Start program will not be receiving any intervention.

INTERVENTIONS:
Behavioral: Healthy Caregivers- Healthy children — The HC2 intervention is an obesity prevention program that provides nutrition and healthy activities programs administered weekly via Zoom or in-person.
  Arms: HC2 intervention Group
Behavioral: Jump Start — The Jump Start intervention is a behavioral health and safety program that provides behavior management and safety programs administered weekly via Zoom or in-person.
  Arms: Jump Start Control Group

SUMMARY:
The purpose of the study is to further develop and examine the Health Caregivers Healthy Children (HC2) program, which encourages obesity prevention through promoting healthy eating and physical activity.

ELIGIBILITY:
Center Inclusion Criteria:

1. have >30 children ages 2-to-5 with a with or at-risk for a disability or special healthcare need
2. Serve low income families
3. Reflect the ethnic diversity of the Miami Dade county Public School System (60% Hispanic, 20% non-Hispanic Black, 20% Non Hispanic White).

Child inclusion criteria:

1. Children with an Individual Education Plan or at-risk based on social and economic variables
2. child ages 2-5
3. child enrolled in a childcare center

Exclusion Criteria:

1) Children with feeding tubes or those that bring their own meals due to dietary restrictions

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index Percentile | Baseline, Up to 3 years
  Body mass index will be collected on children enrolled using participant's height and weight using a percentile score from 0-100
Change in Environment and Policy Assessment and Observation tool) and the Healthy Environment Rating Scale | Baseline, Up to 3 years
  Environment and Policy Assessment and Observation Tool has a total score ranging from 0-100 with the higher score indicating greater quality of nutrition

SECONDARY OUTCOMES:
Change in Healthy Caregivers-Healthy Children (HC2) Survey | Baseline, Up to 3 years
  Teacher and parents complete this survey on the number of reported nutrition and physical activity practices
Change in Health Environment Rating Scale | Baseline, Up to 3 years
  The Healthy Environment Rating Scale has a total score ranging from 0-100 with the higher score indicating increased healthy practices
Change in Parent Stress Index | Baseline, Up to 3 years
  Parents will complete this survey of stress. The Parent Stress Index ranges from 0-100 with higher scores indicating higher levels of stress.
Change in Childcare Worker Job Stress Index | Baseline, Up to 3 years
  The Childcare Worker Job Stress Index is a total score that ranges from 22 to 110 with higher scores indicating higher levels of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Natale, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No